CLINICAL TRIAL: NCT06185036
Title: Histological Validation of dGEMRIC Indices as a Quantitative Biomarker for Cartilage Damage in the Hip Joint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01313; 320030_205091 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cartilage Damage; Osteoarthritis, Hip
Keywords: dGEMRIC; Biomarker
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fixed osteochondral samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators seek to validate 3D model-based dGEMRIC (delayed gadolinium enhanced MRI of cartilage) values against histologic grading of cartilage quality, using osteochondral samples of the femoral head collected during hip replacement surgery.

DETAILED DESCRIPTION:
For patients with advanced hip joint degeneration visible on pelvic radiographs, joint-preserving surgery is often not an option, making joint replacement the primary treatment choice. However, for those with moderate signs of degeneration, the choice between joint-preserving surgery and replacement can be challenging. This decision often relies on imaging techniques such as preoperative direct MR arthrography.

Recent developments in medical imaging have led to new biochemical MRI sequences, such as dGEMRIC. These sequences are valuable for assessing the condition of cartilage before significant morphologic changes occur. By measuring glycosaminoglycan (GAG) content in cartilage, dGEMRIC provides early insight into cartilage degradation. Incorporating these sequences into standard MRI protocols allows the generation of dGEMRIC indices and the creation of 3D models of hip cartilage, improving the overall assessment of the hip joint.

The purpose of this study is to validate 3D model-based dGEMRIC values by comparing them to histologic assessments of cartilage degeneration. The hypothesis is that the dGEMRIC indices from the 3D MRI model will correlate with the histologic grading of cartilage quality in femoral cartilage samples obtained during hip replacement surgery.

This study aims to enroll 25 patients scheduled for total hip arthroplasty. Each participant will undergo preoperative biplanar hip radiographs and direct MR arthrography at 3 Tesla, including the dGEMRIC sequence, according the hospital's standard protocol.

Surgeries will performed by an experienced orthopaedic hip surgeon. The procedure will involve the femoral neck osteotomy, followed by the removal of the head-neck fragment, and the implantation of the hip prosthesis. Osteochondral samples will be taken from four areas of the femoral head. These will be analyzed using toluidine blue and safranin-O staining to assess cartilage damage.

A validated artificial intelligence algorithm will be used for 3D segmentation, visualization and calculation of morphological and biochemical parameters, which will be compared with histological results to determine a dGEMRIC threshold for identifying cartilage damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced hip osteoarthritis.
* Preoperative hip MRI including biochemical sequence (MP2RAGE).
* Indication for hip replacement.

Exclusion Criteria:

* Patients without informed consent.
* Age under 18 years.
* Insufficient language understanding in German, French, or English.
* Previous hip surgeries.
* Neoplastic and inflammatory comorbidities of the hip.
* Post-traumatic or pediatric deformities.
* Avascular necrosis of the femoral head.
* Inadequate MRI image quality (motion artifacts, extra-articular contrast media administration, delay (>45 minutes) between contrast injection and MRI imaging).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the outpatient clinic who meet the inclusion criteria will be informed about the study during orthopaedic consultations. Screening is not required as all necessary information is available from standard diagnostics. Patients will be provided with study and surgical consent forms to be signed after an informed consent interview with one of the investigators. There is no financial compensation for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient of dGEMRIC indices and histological cartilage quality | Within 12 months after histological analysis
  Linear regression analysis will be performed to assess the correlation between dGEMRIC scores and the histological evaluation of cartilage quality.

SECONDARY OUTCOMES:
dGEMRIC indices from 3D MRI cartilage model (T1 relaxation time in milliseconds) | Within 12 months after MRI/patient enrollment
  A validated artificial intelligence based algorithm will be used for automated segmentation and visualization of 3D cartilage models and calculation of dGMERIC values. These dGEMRIC values are displayed topographically and color-coded in the 3D model. This allows visual and three-dimensional assessment of cartilage quality.
Intensity of Toluidine blue staining as a histological value of cartilage damage (Mankin grading 0-14) | Within 1-2 weeks after sample acquisition
  One of the two osteochondral samples from each of the four regions of the femoral head will be fixed for toluidine blue staining to determine the Mankin score. This staining method is used to grade cartilage damage. An experienced histopathologist will evaluate these sections, performing the Mankin grading, which ranges from 0 (indicating no histologic cartilage damage) to 14 (signifying end-stage cartilage damage).
Intensity of Safranin-O staining as a histological value of cartilage damage (Relative red fraction of the RGB scale, 0-255) | Within 1-2 weeks after sample acquisition
  The other osteochondral sample from each region will be used for the Safranin-O staining. An image analysis software (ImageJ, National Institute of Health, Bethesda Md) will be used to quantify the intensity of the Safranin-O staining. This quantification is represented by the relative amount of red in RGB analysis, with intensity values ranging from 0 to 255. This analysis will be performed without reference to the MRI images to ensure objectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Simon D. Steppacher, PD Dr., Principal Investigator — University Hospital of Bern (Inselspital)
Locations (1):
- University Hospital of Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No